CLINICAL TRIAL: NCT01373775
Title: Risk Factors of the Revisit of the Adult Heart Failure Patients in Emergency Department in Siriraj Hospital: The One Year Period.
Brief Title: Risk Factors of the Revisit of the Adult Heart Failure Patients in Emergency Department Siriraj Hospital
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Dr. Phuriphong Songarj, Department of Anesthesiology
Other Study IDs: 740/2551(EC1)
Record Dates: First submitted 2011-06-09; First posted 2011-06-15 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Congestive Heart Failure; Renal Insufficiency
Keywords: Heart failure; Revisit; Emergency room
MeSH Terms: conditions — Heart Failure; Renal Insufficiency; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Revisit: HF patients who revisit the emergency department before the next appointment date.
  Interventions: Other: Patient charts reviewing
- Non-revisit: HF patients who follow up on the appointment date.
  Interventions: Other: Patient charts reviewing

INTERVENTIONS:
Other: Patient charts reviewing — Reviewing chart and identifying risk factors

SUMMARY:
To identify the risk factors of the revisit of the adult HF patients in emergency department.

DETAILED DESCRIPTION:
Because heart failure (HF) is the leading cause of hospitalization and readmission in many hospitals worldwide.

Identifying the risk factors of these HF patients in emergency department is the important reason for the proper management of the HF patients in the future. And can reduce number of hospitalization and readmission in our hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients age from 18 years old
* Patients who were diagnosed HF by the Framingham's criteria10
* Patients who were discharged home from emergency department

Exclusion Criteria:

* Patients age less than 18 years old
* Patients who not met Framingham's criteria, needed hospital admission, were referred to other hospital, and death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical records of 533 patients,who visited the emergency department with the diagnosis of HF (ICD-10 I500, I501 and I509) in the period from 1st Jan 2008 to 31st Dec 2008, were reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 533 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Number of HF patients who were revisited emergency department before the appointment date. | 1 year
  All HF-peatient charts were reviewed and divided in revisit group and non revisit group.

SECONDARY OUTCOMES:
Characteristics of the patients in revisit group | 1 year
  The Characteristics of the patients in both groups such as underlying diseases, ejection fraction, and time for treating in emergency department. The results were compared to find the relation between both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Phuriphong Songarj, MD, Principal Investigator — Department of Anesthesiology
Locations (1):
- Emergency department, Siriraj hospital, Bangkok, Thailand